CLINICAL TRIAL: NCT04899843
Title: Effectiveness of Zinc Supplementation With Topical Retinoids in Acne Vulgaris Patients: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effectiveness of Zinc Supplementation With Topical Retinoids in Acne Vulgaris Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Humayra Rumu, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2021/3959
Record Dates: First submitted 2021-05-11; First posted 2021-05-25 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Acne Vulgaris
Keywords: AV Zinc GAGS Serum zinc level
MeSH Terms: conditions — Acne Vulgaris | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: Newly diagnosed Acne vulgaris patients
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): This arm includes 61 acne vulgaris patients receiving topical retinoids
  Interventions: Dietary Supplement: Zinc sulphate tablet 20 mg
- Control (Placebo Comparator): This arm includes 61 acne vulgaris patients receiving topical retinoids
  Interventions: Dietary Supplement: Placebo tablet 20 mg

INTERVENTIONS:
Dietary Supplement: Zinc sulphate tablet 20 mg — Zinc sulphate tablet 20 mg daily orally for 8 weeks along with topical retinoids.
  Arms: Experimental
Dietary Supplement: Placebo tablet 20 mg — Placebo tablet 20 mg daily orally for 8 weeks along with topical retinoids
  Arms: Control

SUMMARY:
The study was 8 weeks, randomized, double-blind, placebo-controlled trial to assess the effect of zinc sulphate on symptoms of mild and moderate acne vulgaris in 122 patients. Participants was assessed at baseline, and 8 weeks. Subjects was randomized to receive either 20 mg elemental zinc daily or 20 mg placebo tablet daily for 8 weeks. The primary outcome was the measure of the GAGS score and the secondary measure includes serum zinc level and evaluate adverse effects.

DETAILED DESCRIPTION:
Acne vulgaris (AV) is the eighth most prevalent disease worldwide. Acne is a self-limiting condition, it may cause significant psychological and social problems, depression, disfigurement, and scarring that can persist for a lifetime. Multiple factors contribute to acne pathogenesis including increased sebum production, aberrant keratinization of the pilosebaceous duct, bacteria such as Propionibacterium acnes, hormonal influences, the skin microbiome, and chronic inflammation. Relapse rates in patients with acne after treatment with standard of care vary between 10% and 60%. Recent trials attempted to assess the effect of zinc in reducing the severity of symptoms of acne vulgaris patients. This study evaluates whether there is any role of zinc in reducing acne symptoms between those who did and did not receive zinc in an 8 weeks period. This includes 122 acne vulgaris patients who were recruited from Dermatology and Venereology OPD of BSMMU. Participants took either 20 mg elemental zinc daily in the form of zinc sulphate tablet or 20 mg placebo tablet daily for 8 weeks. Initially, baseline serum zinc level was measured and repeated again after 8 weeks of intervention. A baseline acne symptoms survey was done by GAGS score and also repeated at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed mild and moderate AV patients diagnosed by a dermatologist at the outpatient Department of Dermatology and Venereology,
* Age: 11-35 years,
* Gender: Both male and female

Exclusion Criteria:

* Pregnancy and lactation,
* History of oral contraceptive pills, zinc, and iron intake,
* Suffering from any cosmetic induced acne

Ages: 11 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Acne vulgaris severity score assessment | 8 weeks
  Assess the severity score of acne vulgaris symptoms by GAGS(Global Acne Grading System) at baseline, and after 8 weeks.
  And compare the score between two groups. GAGS scores : 1-18 Mild, 19-30 Moderate

SECONDARY OUTCOMES:
Biochemical assessment and evaluate the adverse effects | 8 weeks
  Serum zinc level was assessed at baseline and after 8 weeks intervention.Compare the serum zinc level between two group. Adverse effects are evaluated which reported by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Md. Sayedur Rahman, MBBS, Mphil, FCPS, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Basic Science and Paraclinical Science of BSMMU, Dhaka, Bangladesh